CLINICAL TRIAL: NCT05591170
Title: The Effect of Single High Dose of Vitamin D on Serum Levels of Its Metabolites
Brief Title: Effect of Single High Dose of Cholecalciferol on Serum Metabolites of Vitamin D
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Department of Endocrinology, Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Dorota Lesczyńska, MD, Department of Endocrinology, Centre of Postgraduate Medical Education
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 042021082021
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin D; 25(OH)D3; 25(OH)D2; 3-epi-25(OH)D3; 24,25(OH)2D3; 1,25(OH)2D3
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group (Experimental): Participants received single, high, oral dose of vitamin D3 (120,000 IU), serum 25(OH)D3, 25(OH)D2, 24,25(OH)2D3, 3-epi-25(OH)D3, 1,25(OH)2D3, 24,25(OH)2D3/25(OH)D3 ratio, and 25(OH)D3/3-epi-25(OH)D3 ratio concentration (measured by LC-MS/MS) at baseline, 3 days and 7 days after bolus dose were measured.
  The percentage of fat tissue was determined using Dual-Energy X-Ray Absorptiometry (DXA).
  Interventions: Drug: Cholecalciferol 120 000 IU
- Control Group (No Intervention): Serum 25(OH)D3, 25(OH)D2, 24,25(OH)2D3, 3-epi-25(OH)D3, 1,25(OH)2D3, 24,25(OH)2D3/25(OH)D3 ratio, and 25(OH)D3/3-epi-25(OH)D3 ratio concentration (measured by LC-MS/MS) were measured at baseline, 3 days and 7 days after.
  The percentage of fat tissue was determined using Dual-Energy X-Ray Absorptiometry (DXA).

INTERVENTIONS:
Drug: Cholecalciferol 120 000 IU — single, oral administration of high dose of vitamin D
  Other Names: Solderol
  Arms: Study Group

SUMMARY:
The aim of this interventional study is to assess the effect of the single high dose of vitamin D on its serum metabolites in elderly.

The main questions it attempts to answer is:

1. what is the effect of a single, high, oral dose of vitamin D3 (120,000 IU) on serum 25(OH)D3, 25(OH)D2, 24,25(OH)2D3, 3-epi-25(OH)D3, 1,25(OH)2D3, 24,25(OH)2D3/25(OH)D3 ratio, and 25(OH)D3/3-epi-25(OH)D3 ratio concentration at baseline, 3 days and 7 days after administration, compared to control group.
2. what is the influence of percentage of fat tissue on serum metabolites of vitamin D and their changes after bolus dose, compared to control group.

DETAILED DESCRIPTION:
Vitamin D belongs to dietary micronutriens and it is known for pleiotropic actions, going far beyond its classical function of maintenance of calcium/phosphorous homeostasis. The extra-skeletal effects of vitamin D include the role in cellular proliferation, differentiation, and immune modulation. Therefore, vitamin D has become the subject of numerous studies in relation to its potential protective effect in pathophysiology of diabetes, cardiovascular diseases, autoimmune diseases, infections and cancer.

The most common form of vitamin D is 25(OH)D3 - it can be obtained by photochemical reaction in the skin and through diet via animal-based food. 25(OH)D2 may be found in some plant-based food and has lower affinity to vitamin D binding protein, therefore it has a shorter half-life in the blood. In many countries, due to insufficient skin synthesis, vitamin D has to be acquired through fortified food and supplements in different dosing schedules (e.g. once daily, once weekly). Higher doses of vitamin D taken less frequently may significantly improve patients' adherence to recommended treatment regimens. However, there are arising questions about the efficacy and safety of such interventions. 1,25(OH)2D3 is the product of 1-hydroxylation of 25(OH)D3 in kidneys and it is the active form of vitamin D with a short half-life in the blood, while 24,25(OH)2D3 is the product of the reaction of 24-hydroxylase and it is considered inactive. The measurement of serum levels of both metabolites may contribute to better understanding the mechanisms protecting against too high increase of active forms of vitamin D.

In the study, the investigators aim to establish the changes of serum vitamin D metabolites (namely 25OHD, 25(OH)D3, 24,25(OH)2D3, 25(OH)D2, 3-epi-25(OH)D3 and 1,25(OH)2D3) and chosen ratios after oral administration of 120 000 IU of vitamin D 3 days and 7 days after the intervention in hospitalized elderly patients. The investigators also address a question if the change of serum vitamin D metabolites after single high dose of vitamin D3 is dependent on the body fat percentage and severity of vitamin D deficiency. Quantitative analyses were performed using liquid chromatography with tandem mass spectrometry (LC-MS/MS).

ELIGIBILITY:
Inclusion Criteria:

* written, informed consent,
* age ≥ 60 years-old,
* admission to the hospital due to emergency reasons.

Exclusion Criteria:

* hypercalcemia,
* nephrolithiasis,
* kidney insufficiency,
* documented vitamin D3 metabolism disorders such as sarcoidosis, parathyroid disease or genetic defects,
* vitamin D3 supplementation within 6 months prior to the hospitalisation.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Changes of serum vitamin D metabolites after the administration of 120 000 IU cholecalciferol compared to control group. | Measurements at baseline, 3 days and 7 days after.
  Changes of serum 25(OH)D3, 25(OH)D2, 24,25(OH)2D3, 3-epi-25(OH)D3, 1,25(OH)2D3, 24,25(OH)2D3/25(OH)D3 ratio, and 25(OH)D3/3-epi-25(OH)D3 ratio concentration at baseline, 3 days and 7 days after the intervention, compared to control group.

SECONDARY OUTCOMES:
Influence of percentage of fat tissue on serum concentration of metabolites of vitamin D and their changes after bolus dose. | Dual-Energy X-Ray Absorptiometry (DXA) at baseline, measurements of vitamin D metabolites at baseline, 3 days and 7 days after.
  Influence of percentage of fat tissue on serum 25(OH)D3, 25(OH)D2, 24,25(OH)2D3, 3-epi-25(OH)D3, 1,25(OH)2D3 and their changes at baseline, 3 days and 7 days after the intervention, compared to control group.

CONTACTS AND LOCATIONS:
Overall Officials: Wojciech Zgliczyński, Prof., Study Chair — Department of Endocrinology, Centre of Postgraduate Medical Education
Locations (1):
- Department of Endocrinology, Centre of Postgraduate Medical Education, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ilahi M, Armas LA, Heaney RP. Pharmacokinetics of a single, large dose of cholecalciferol. Am J Clin Nutr. 2008 Mar;87(3):688-91. doi: 10.1093/ajcn/87.3.688. PMID 18326608
- [Background] Saleh L, Tang J, Gawinecka J, Boesch L, Fraser WD, von Eckardstein A, Nowak A. Impact of a single oral dose of 100,000 IU vitamin D3 on profiles of serum 25(OH)D3 and its metabolites 24,25(OH)2D3, 3-epi-25(OH)D3, and 1,25(OH)2D3 in adults with vitamin D insufficiency. Clin Chem Lab Med. 2017 Oct 26;55(12):1912-1921. doi: 10.1515/cclm-2016-1129. PMID 28328526
- [Derived] Leszczynska D, Szatko A, Kowalski K, Raczkiewicz D, Ostrowska M, Misiorowski W, Zgliczynski W, Glinicki P. The Effect of a Single High Dose of Vitamin D on Serum Levels of Its Metabolites in the Elderly. Front Biosci (Landmark Ed). 2022 Oct 25;27(10):289. doi: 10.31083/j.fbl2710289. PMID 36336861